CLINICAL TRIAL: NCT04050826
Title: An Exploratory Study in Healthy Volunteers to Identify Factors Influencing Bioequivalence Studies on Moderately Lipophilic Drugs Using Dermal Open Flow Microperfusion (dOFM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDA02_AIM2_Main
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Healthy; Dermal Pharmacokinetic Measurements
Keywords: Dermal open flow microperfusion
MeSH Terms: interventions — Lidocaine; Prilocaine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dermal Pharmacokinetic study (Experimental): Measurement of dermal pharmacokinetic (PK) parameter (AUC, Cmax) of lidocaine/ prilocaine using dOFM after topical application of three lidocaine/prilocaine products in 20 participants.
  After baseline sampling (1 hour pre-dose) the three lidocaine/prilocaine products will be applied and removed after 3 hours. ISF and blood sampling will be continued for a duration of 12 hours post-dose. Additionally different physical parameters (e.g. TEWL) will be measured.
  Interventions: Drug: Lidocaine 2.5% and Prilocaine 2.5% cream, USP (Actavis Pharma incorporated, USA); Drug: Lidocaine 2.5% and Prilocaine 2.5% cream (E. Fougera & Co. a division of Fougera Pharmaceuticals Inc., USA); Drug: Oraqix Parodontal-Gel (Dentsply Detrey GmbH, Germany); Device: Dermal open flow microperfusion; Procedure: Blood sampling

INTERVENTIONS:
Drug: Lidocaine 2.5% and Prilocaine 2.5% cream, USP (Actavis Pharma incorporated, USA) — Topical application
  Other Names: Reference product
Drug: Lidocaine 2.5% and Prilocaine 2.5% cream (E. Fougera & Co. a division of Fougera Pharmaceuticals Inc., USA) — Topical application
  Other Names: Generic test product
Drug: Oraqix Parodontal-Gel (Dentsply Detrey GmbH, Germany) — Topical application
  Other Names: Non-equivalent test product
Device: Dermal open flow microperfusion — Dermal open flow microperfusion will be used to collect interstitial fluid in order to assess lidocaine/prilocaine concentration in the dermis.
  16 dOFM probes will be implanted per participant (8 test-sites; 2 dOFM probes per test-site).
  From each dOFM probe 13 samples will be taken (1 pre-dose, 12 post-dose).
Procedure: Blood sampling — 1 sample will be taken pre-dose and 12 samples post-dose.

SUMMARY:
The overall aim of this clinical study is to develop a general bioequivalence (BE) testing method using dermal open flow microperfusion (dOFM) for dermatological drug products. In this study BE of different lidocaine/prilocaine products will be assessed and factors that influence dOFM data variability will be evaluated.

DETAILED DESCRIPTION:
The study will involve 20 healthy adult participants. Dermal pharmacokinetic (PK) profile of three different lidocaine/prilocaine products will be assessed in parallel at different skin sites on the same participant.

For BE evaluations a reference product will be compared against itself and an approved generic test product as positive control and against a non-equivalent test product as negative control. Additionally different non-invasive measurements (e.g. TEWL) will be conducted and results will be correlated with lidocaine/prilocaine PK data to identify factors that might influence skin penetration.

dOFM probes will be inserted into the dermis to monitor the dermal drug concentrations up to 12 h post-dose in topically treated skin sites. Blood samples will be drawn to rule out systemic appearance of lidocaine and/or prilocaine.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years inclusive.
2. Males and/or non-pregnant, non-breast feeding females (subjects need to be informed about adequate contraceptive methods).
3. Able to read, understand, and sign the written informed consent form.
4. Willing to follow the protocol requirements and comply with protocol restrictions.

Exclusion Criteria:

1. Social Habits

   1. Smoker who is not willing to restrain from smoking during the in-house visit (Visit 2).
   2. History of drug and/or alcohol abuse within one year of start of study as judged by the investigator.
2. Medications: Current treatment with systemically effective corticosteroids, monoamine oxidase (MAO) inhibitors, systemic non-selective beta-blockers, warfarin or anticholinergic drugs, or use of any medications referred in the prescription information of the products. Hormonal contraceptive or hormone replacement therapy, routine vitamins or other prescribed medication are allowed if dose is stable.
3. Diseases

   1. Congenital or idiopathic methemoglobinemia
   2. History of deep vein thrombosis (DVT)/pulmonary emboly (PE)
   3. Inherited blood disorders (such as factor V Leiden) who are prone to hypercoagulable state
   4. Glucose-6-phosphate dehydrogenase deficiencies
   5. Presence of any acute or chronic diseases or malignancies unless deemed not clinically significant by the investigator.
4. Any reason which, in the opinion of the investigator, would prevent the subject from safely participating in the study.
5. Any abnormalities found at physical examination or vital signs, unless deemed not clinically significant by the investigator.
6. Clinically significant abnormal laboratory evaluation results, as deemed by the investigator.
7. Clinically significant abnormal 12-lead ECG at screening, as deemed by the investigator.
8. Positive results to the test for hepatitis B antigen or hepatitis C antibodies.
9. Positive HIV test.
10. Positive alcohol breath test.
11. Blood donation within 30 days or significant loss of blood or plasma (more than 550 ml) within 90 days prior to screening.
12. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
13. Any food allergy, intolerance, restriction or special diet that, in the opinion of the investigator, could contraindicate the subject's participation in this study.
14. Known or suspected allergy/hypersensitivity to lidocaine or prilocaine, known history of sensitivity to local anesthetics of the amide type or to any other component of the product, other related products, or any inactive ingredients.
15. Tattoos or broken and/or damaged skin at the application areas.
16. Active skin diseases like psoriasis or atopic dermatitis, as judged by the investigator.
17. Scarring at the anterior part of the thighs.
18. Subjects prone to keloid or hypertrophic scar formation or any known wound healing disorder.
19. Recent and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.), as judged by the investigator.
20. Not willing to avoid excessive sun exposure, steam baths, sauna, swimming and other strenuous activities between Visit 2 and the end-of-study examination to ensure good tissue regeneration.
21. Not willing to refrain from shaving the anterior of the thighs or using skin care products on the anterior of the thighs for at least 5 days prior to start of Visit 2.
22. Pronounced hairiness on the thighs that may negatively affect BE testing.
23. Known allergy/hypersensitivity to any of the materials/supplies used during the study.
24. Presence of needle phobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Area under the dermal concentration versus time curve for lidocaine | 13 hours
  Dermal concentrations (ng/mL) of lidocaine will be measured to calculate the area under the dermal concentration versus time curve AUC (ng*h/mL).
Area under the dermal concentration versus time curve for prilocaine | 13 hours
  Dermal concentrations (ng/mL) of prilocaine will be measured to calculate the area under the dermal concentration versus time curve AUC (ng*h/mL).
Maximal dermal concentration of lidocaine | 13 hours
  Dermal concentrations (ng/mL) of lidocaine will be measured to calculate the maximal dermal concentration (ng/mL).
Maximal dermal concentration of prilocaine | 13 hours
  Dermal concentrations (ng/mL) of prilocaine will be measured to calculate the maximal dermal concentration (ng/mL).

SECONDARY OUTCOMES:
Blood lidocaine concentrations versus time curve | 13 hours
  Lidocaine concentrations (ng/mL) in the blood will be measured to obtain the concentration-time curves in the blood.
Blood prilocaine concentrations versus time curve | 13 hours
  Prilocaine concentrations (ng/mL) in the blood will be measured to obtain the concentration-time curves in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- CTU - Clinical Trials Unit, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodenlenz M, Tiffner KI, Raml R, Augustin T, Dragatin C, Birngruber T, Schimek D, Schwagerle G, Pieber TR, Raney SG, Kanfer I, Sinner F. Open Flow Microperfusion as a Dermal Pharmacokinetic Approach to Evaluate Topical Bioequivalence. Clin Pharmacokinet. 2017 Jan;56(1):91-98. doi: 10.1007/s40262-016-0442-z. PMID 27539717
- [Background] Bodenlenz M, Dragatin C, Liebenberger L, Tschapeller B, Boulgaropoulos B, Augustin T, Raml R, Gatschelhofer C, Wagner N, Benkali K, Rony F, Pieber T, Sinner F. Kinetics of Clobetasol-17-Propionate in Psoriatic Lesional and Non-Lesional Skin Assessed by Dermal Open Flow Microperfusion with Time and Space Resolution. Pharm Res. 2016 Sep;33(9):2229-38. doi: 10.1007/s11095-016-1960-y. Epub 2016 Jun 6. PMID 27271272
- [Background] Bodenlenz M, Aigner B, Dragatin C, Liebenberger L, Zahiragic S, Hofferer C, Birngruber T, Priedl J, Feichtner F, Schaupp L, Korsatko S, Ratzer M, Magnes C, Pieber TR, Sinner F. Clinical applicability of dOFM devices for dermal sampling. Skin Res Technol. 2013 Nov;19(4):474-83. doi: 10.1111/srt.12071. Epub 2013 Apr 13. PMID 23581539
- [Background] Dragatin C, Polus F, Bodenlenz M, Calonder C, Aigner B, Tiffner KI, Mader JK, Ratzer M, Woessner R, Pieber TR, Cheng Y, Loesche C, Sinner F, Bruin G. Secukinumab distributes into dermal interstitial fluid of psoriasis patients as demonstrated by open flow microperfusion. Exp Dermatol. 2016 Feb;25(2):157-9. doi: 10.1111/exd.12863. Epub 2015 Nov 23. No abstract available. PMID 26439798
- [Background] Tiffner K, Boulgaropoulos B, Hofferer C, Birngruber T, Porksen N, Linnebjerg H, Garhyan P, Lam ECQ, Knadler MP, Pieber TR, Sinner F. Quantification of Basal Insulin Peglispro and Human Insulin in Adipose Tissue Interstitial Fluid by Open-Flow Microperfusion. Diabetes Technol Ther. 2017 May;19(5):305-314. doi: 10.1089/dia.2016.0384. Epub 2017 Mar 22. PMID 28328234
- See also: In Vivo Dermal Open Flow Microperfusion: A Novel Approach to Evaluating Topical Bioavailability and Bioequivalence — https://www.fda.gov/downloads/Drugs/NewsEvents/UCM591892.pdf